CLINICAL TRIAL: NCT07315854
Title: A Prospective, Single-Center, Exploratory Phase II Clinical Study of Iparomlimab and Tuvonralimab (QL1706) Combined With Chemotherapy in the Treatment of Previously Untreated Advanced or Metastatic Gastric or Gastroesophageal Junction Cancer
Brief Title: Iparomlimab and Tuvonralimab (QL1706) Combined With Chemotherapy for Previously Untreated Advanced or Metastatic Gastric or Gastroesophageal Junction Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, dengwei, Chief Physician, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BFHHS20250012; BFHHS20250012 (Registry Identifier: Beijing Friendship Hospital, Capital Medical University)
Record Dates: First submitted 2025-12-20; First posted 2026-01-02 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Gastric Cancer (GC); Gastroesophageal Junction Cancer; Advanced Gastric Cancer; Metastatic Gastric Cancer
Keywords: Iparomlimab and Tuvonralimab; QL1706; Advanced or Metastatic Gastric Cancer; PD-1/CTLA-4 Bispecific Antibody; Immunotherapy; Chemotherapy Combination; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QL1706 + SOX (Experimental): Participants will receive induction therapy with Iparomlimab and Tuvonralimab (QL1706) combined with SOX chemotherapy (Oxaliplatin and S-1) for 6 cycles (every 3 weeks). This is followed by maintenance therapy with QL1706 and S-1 until disease progression, intolerable toxicity, or other discontinuation criteria are met.
  Interventions: Drug: Iparomlimab and Tuvonralimab (QL1706); Drug: SOX Chemotherapy

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab (QL1706) — Administered via intravenous (IV) infusion at a dose of 5 mg/kg on Day 1 of each 3-week cycle.
Drug: SOX Chemotherapy — Oxaliplatin: 130mg/m2, iv.gtt, single infusion, 21 days as a cycle, Day 1. Tigio: 40mg (body surface area(BSA)<1.25m2), 50mg (BSA≥1.25m2, and BAS<1.5m2), 60mg (BSA ≥1.5m2), p.o, bid, 21 days as a cycle, Day 1-14.

SUMMARY:
The goal of this Phase II clinical trial is to evaluate the efficacy and safety of Iparomlimab and Tuvonralimab (QL1706) combined with SOX chemotherapy (S-1 plus Oxaliplatin) in patients with previously untreated advanced or metastatic gastric cancer or gastroesophageal junction cancer.

The main questions it aims to answer are:

1、What is the objective response rate (ORR) of the combination of QL1706 and SOX chemotherapy? 2、What are the safety and tolerability of this combination therapy? Participants will：

1. Receive Iparomlimab and Tuvonralimab (QL1706) via intravenous infusion every 3 weeks.
2. Receive SOX chemotherapy (Oxaliplatin via intravenous infusion on Day 1 and S-1 orally twice daily for 14 days) every 3 weeks for up to 6 cycles.
3. Continue maintenance therapy with QL1706 combined with S-1 after 6 cycles until disease progression or unacceptable toxicity.
4. Undergo tumor imaging assessments (CT or MRI) every 6 weeks for the first 24 weeks, and then every 9 weeks thereafter to monitor the disease.

DETAILED DESCRIPTION:
Study Design: This is a prospective, single-center, single-arm, exploratory Phase II clinical study designed to evaluate the efficacy and safety of Iparomlimab and Tuvonralimab (QL1706) combined with SOX chemotherapy (S-1 and Oxaliplatin) as a first-line treatment for patients with advanced or metastatic gastric or gastroesophageal junction (GEJ) cancer. The study aims to enroll approximately 32 eligible participants.

Intervention and Treatment Regimen: Eligible participants will undergo a screening period of up to 3 weeks. Upon enrollment, subjects will receive the combination therapy in 3-week cycles as follows:

Induction Phase (Cycles 1-6):

Iparomlimab and Tuvonralimab (QL1706): Administered intravenously at a fixed dose of 5 mg/kg on Day 1 of each cycle.

Oxaliplatin: Administered intravenously at a dose of 130 mg/m² on Day 1 of each cycle.

S-1 (Tegafur, Gimeracil, Oteracil): Administered orally twice daily (after breakfast and dinner) on Days 1-14, followed by a 7-day rest period. The dose is calculated based on body surface area (BSA): 40 mg/dose for BSA ≤1.25 m²; 50 mg/dose for BSA 1.25-1.5 m²; and 60 mg/dose for BSA >1.5 m².

Maintenance Phase (Cycle 7 onwards):

After completing 6 cycles of the combination therapy, patients without disease progression or intolerable toxicity will continue with maintenance therapy consisting of QL1706 (5 mg/kg IV q3w) combined with S-1 (oral, same schedule) until disease progression, death, intolerable toxicity, or withdrawal of consent. Note: Oxaliplatin is discontinued in the maintenance phase.

Assessments: Efficacy is assessed using tumor imaging (CT/MRI) according to RECIST v1.1 criteria. Tumor assessments are performed every 6 weeks for the first 24 weeks and every 9 weeks thereafter. The primary endpoint is the Objective Response Rate (ORR). Secondary endpoints include Disease Control Rate (DCR), Progression-Free Survival (PFS), Overall Survival (OS), and 1-year PFS/OS rates. Safety is monitored throughout the study via adverse event reporting (NCI-CTCAE v5.0), laboratory tests, and physical examinations.

Follow-up: After treatment discontinuation, patients will enter a safety follow-up period (90 days post-last dose) and a survival follow-up period, where survival status and subsequent anti-tumor therapies will be collected every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in the clinical study; fully understand and are informed about the study and sign the Informed Consent Form (ICF); willing to follow and able to complete all trial procedures.
* Age 18-80 years, gender is not limited.
* Patients with locally advanced unresectable, recurrent unresectable, or metastatic gastric cancer (GC) or gastroesophageal junction cancer (GEJC) confirmed by imaging and other examinations, and histopathologically confirmed as adenocarcinoma.
* Provide a report confirming HER2 overexpression or amplification negativity; defined as IHC 0/1+, or IHC 2+ with FISH/ISH negative.
* No prior systemic therapy for advanced or metastatic GC/GEJC (including anti-HER-2 therapy). Patients who have received adjuvant or neoadjuvant therapy (including chemotherapy, radiotherapy, or chemoradiotherapy) for GC/GEJC are eligible if the time to first recurrence or disease progression is greater than 6 months from the end of the last treatment. Prior use of anti-tumor Traditional Chinese Medicine preparations is allowed but must be discontinued at least 2 weeks before enrollment.
* ECOG performance status score of 0 or 1.
* Must have at least one measurable lesion according to RECIST v1.1 definitions.
* All acute toxicities caused by prior anti-tumor therapy or surgery must have resolved to Grade 0-1 (according to NCI CTCAE v5.0) or to the level specified in the inclusion/exclusion criteria. Alopecia, fatigue, and hearing loss, or other toxicities considered by the investigator not to pose a safety risk to the subject, are excluded.
* Adequate organ function (laboratory tests within 7 days prior to treatment):

  * Hematology (No blood transfusion, G-CSF use, or drug correction within 14 days prior to screening):
  * White blood cell count (WBC) ≥ 3,000/mm³ (3.0 × 10⁹/L);
  * Absolute neutrophil count (ANC) ≥ 1,500/mm³ (1.5 × 10⁹/L);
  * Platelet count (PLT) ≥ 100,000/mm³ (100 × 10⁹/L);
  * Hemoglobin (Hb) ≥ 9.0 g/dL (90 g/L).
* Biochemistry (No albumin transfusion within 14 days prior to screening):

  * Albumin ≥ 3.0 g/dL (30 g/L);
  * Creatinine ≤ 1.5 × Upper Limit of Normal (ULN) or Creatinine Clearance ≥ 50 ml/min (calculated using the Cockcroft-Gault formula);
  * Total Bilirubin (BIL) ≤ 1.5 × ULN;
  * Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) levels ≤ 2.5 × ULN; for patients with liver metastases, ≤ 5 × ULN.
* Coagulation: International Normalized Ratio (INR) ≤ 1.5, Prothrombin Time (PT), and Activated Partial Thromboplastin Time (APTT) ≤ 1.5 × ULN.
* Urine: Urine protein < 2+; if urine protein is ≥ 2+, 24-hour urine protein quantification must be ≤ 1g.
* Life expectancy ≥ 3 months.
* Women of childbearing potential must undergo a serum or urine pregnancy test within 7 days before starting treatment, with a negative result, and must not be lactating. All enrolled patients must use adequate barrier contraception throughout the treatment cycle and for 6 months after the end of treatment.

Exclusion Criteria:

* Known squamous cell carcinoma, undifferentiated carcinoma, other histological types of gastric cancer, or mixed gastric cancer containing other histological types.
* Active malignant tumors within the past 2 years, other than the tumor under study. Exceptions include subjects with locally curable cancers (that have been cured), such as basal or squamous cell skin cancer, superficial bladder cancer, and carcinoma in situ of the cervix or breast.
* Participation in a study of an investigational drug or receipt of investigational treatment or use of an investigational device within 4 weeks prior to the first dose.
* Enrollment in another clinical study, unless it is an observational, non-interventional clinical study or the follow-up period of an interventional study (defined as >4 weeks since the last dose of the previous clinical study or >5 half-lives of the study drug).
* Untreated Central Nervous System (CNS) metastases, or uncontrolled or symptomatic active CNS metastases. Patients with fully treated CNS metastases may be enrolled if neurological symptoms have returned to baseline levels at least 4 weeks prior to enrollment (excluding residual signs or symptoms related to CNS treatment). Additionally, subjects must have discontinued corticosteroids or be on a stable or tapering dose of prednisone ≤ 10 mg/d (or equivalent dose of other corticosteroids) for at least 4 weeks prior to enrollment.
* Pleural effusion or ascites that remains uncontrolled despite puncture and drainage within 14 days prior to enrollment; symptomatic or moderate-to-large pericardial effusion.
* Weight loss of more than 20% within 2 months prior to enrollment.
* Received the following treatments or medications prior to enrollment:

  * Major surgery within 28 days prior to enrollment (tissue biopsy for diagnosis and PICC/port implantation are allowed).
  * Use of immunosuppressive drugs within 14 days prior to enrollment, excluding nasal/inhaled corticosteroids or physiological doses of systemic steroids (i.e., ≤ 10 mg/d prednisone or equivalent).
  * Vaccination with live attenuated vaccines within 28 days prior to enrollment or planned during the study period and within 60 days after the end of study drug treatment.
  * Local anti-tumor therapy (e.g., radiotherapy or tumor embolization) within 28 days prior to enrollment.
* Diagnosed with any other malignant tumor within 5 years prior to entering the study, except for cured cutaneous basal cell carcinoma or squamous cell carcinoma, superficial bladder cancer, carcinoma in situ of the cervix, ductal carcinoma in situ of the breast, and papillary thyroid carcinoma amenable to local treatment.
* Presence of any active, known, or suspected autoimmune disease. Subjects in a stable state not requiring systemic immunosuppressive therapy are allowed, such as Type I diabetes, hypothyroidism requiring only hormone replacement therapy, and skin diseases not requiring systemic treatment (e.g., vitiligo, psoriasis, alopecia).
* Prior treatment with any anti-PD-1, anti-PD-L1, anti-CTLA-4 antibody, or any other antibody or drug targeting T-cell co-stimulation or checkpoint pathways.
* Significant clinical bleeding symptoms or definite bleeding tendency within 3 months prior to enrollment; gastrointestinal perforation and/or fistula within 6 months prior to enrollment; arterial/venous thromboembolic events within 6 months prior to enrollment, such as cerebrovascular accident (including TIA, cerebral infarction), deep vein thrombosis, and pulmonary embolism (except for those with gastric cancer bleeding/perforation where symptoms disappeared after surgical resection).
* Major vascular disease within 6 months before the start of study treatment (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis).
* Severe, unhealed, or dehisced wounds, active ulcers, or untreated fractures.
* Presence of > Grade 1 peripheral neuropathy.
* History of intestinal obstruction and/or clinical signs or symptoms of gastrointestinal obstruction within 6 months before starting study treatment, including incomplete obstruction related to the underlying disease or requiring routine parenteral hydration, parenteral nutrition, or tube feeding. Patients with incomplete obstruction/obstruction syndrome at initial diagnosis who have symptom relief after definitive (surgical) treatment may be enrolled.
* Interstitial lung disease, non-infectious pneumonitis, or uncontrolled systemic diseases (e.g., diabetes, hypertension, pulmonary fibrosis, acute pneumonia, etc.).
* Known history of active tuberculosis.
* Known allergy to the study drug or any of its excipients; or history of severe allergic reactions to other monoclonal antibodies.
* HIV infection or known Acquired Immunodeficiency Syndrome (AIDS); untreated active hepatitis (Hepatitis B defined as HBV-DNA ≥ 500 IU/ml; Hepatitis C defined as anti-HCV positive and HCV RNA above the lower limit of detection) or co-infection with Hepatitis B and C.
* Poorly controlled clinical cardiac symptoms or diseases, such as: (1) NYHA Class II or higher cardiac insufficiency or LVEF < 50% on echocardiography; (2) Severe/unstable angina; (3) Myocardial infarction within 12 months prior to enrollment; (4) Clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention; (5) Symptomatic congestive heart failure; (6) QTc > 480 ms.
* Systemic use of antibiotics ≥ 7 days within 4 weeks prior to enrollment, or unexplained fever > 38.5°C during screening/before first dose (fever due to tumor causes is allowed per investigator judgment).
* Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
* Participation in any other drug clinical study within 4 weeks or 5 half-lives prior to enrollment.
* Known history of psychotropic drug abuse or drug addiction.
* Presence of other severe physical or mental illnesses or laboratory abnormalities that may increase the risk of participation, interfere with study results, or render the patient unsuitable for the study in the opinion of the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From baseline until disease progression or loss of clinical benefit, assessed every 6 weeks for the first 24 weeks, then every 9 weeks, up to approximately 2 years.
  ORR is defined as the percentage of participants who achieve a Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR), as assessed by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | From baseline until disease progression or loss of clinical benefit, assessed every 6 weeks for the first 24 weeks, then every 9 weeks, up to approximately 2 years.
  DCR is defined as the percentage of participants whose Best Overall Response (BOR) is confirmed as Complete Response (CR), Partial Response (PR), or Stable Disease (SD), as assessed by the investigator according to RECIST v1.1.
Progression-Free Survival (PFS) | From enrollment to the date of first documented progression or death, assessed up to approximately 2 years.
  PFS is defined as the time from the date of enrollment to the date of the first documented disease progression (according to RECIST v1.1) or death from any cause, whichever occurs first.
Overall Survival (OS) | From enrollment to the date of death, assessed up to approximately 2 years.
  OS is defined as the time from the date of enrollment to the date of death due to any cause.
1-Year Progression-Free Survival (PFS) Rate | At 1 year after enrollment.
  The proportion of participants who are alive and free of disease progression at 1 year after enrollment.
1-Year Overall Survival (OS) Rate | At 1 year after enrollment.
  The proportion of participants who are alive at 1 year after enrollment.
Incidence and Severity of Adverse Events (AEs) | From the time of informed consent through 90 days after the last dose of study drug.
  Safety and tolerability will be evaluated by monitoring the incidence and severity of Adverse Events (AEs), Serious Adverse Events (SAEs), Treatment-Related Adverse Events (TRAEs), and Immune-Related Adverse Events (irAEs). Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared publicly. The study protocol emphasizes strict confidentiality of subject data. Aggregate data may be available upon reasonable request to the principal investigator.